CLINICAL TRIAL: NCT02989922
Title: A Randomized Controlled Multicentered Phase 2/3 Study to Evaluate SHR-1210 (PD-1 Antibody) in Subjects With Advanced Hepatocellular Carcinoma (HCC) Who Failed or Intolerable to Prior Systemic Treatment
Brief Title: A Study to Evaluate SHR-1210 in Subjects With Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II/III-HCC
Record Dates: First submitted 2016-11-22; First posted 2016-12-12 (Estimated); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2017-12

CONDITIONS: Hepatocellular Carcinoma Non-Resectable
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHR-1210 Q2W (Experimental): Subjects receive SHR-1210 intravenous at the dose 3mg/kg on Day 1 every 2 weeks
  Interventions: Biological: SHR-1210
- SHR-1210 Q3W (Experimental): Subjects receive SHR-1210 intravenous at the dose 3mg/kg on Day 1 every 3 weeks
  Interventions: Biological: SHR-1210

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody

SUMMARY:
This a randomized controlled Phase 2/3 study to evaluate the efficacy and safety of SHR-1210 in subjects with advanced HCC who failed or intolerable to prior systemic treatment. The primary study hypothesis is that SHR-1210 treatment improves Objective Response Rate and Overall Survival when compare with SOC.

DETAILED DESCRIPTION:
In June 2017, this study was revised to expand the Phase 2 part to enroll more subjects and remove the Phase 3 part under the same protocol. A Phase 3 study will be initiated separately.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HCC in advanced stage; not suitable to surgery or local regional treatment; with at least one measurable lesion per RECIST 1.1
2. Failed or intolerable to at least one prior systemic treatment for advanced HCC
3. ECOG Performance Status of 0 or1
4. Child-Pugh Class A or B with 7 points
5. Life Expectancy of at least 12 weeks
6. HBV DNA<500 IU/ml
7. Adequate organ function
8. Male or female participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 60 days for female subjects and 120 days for male subjects after the last dose of study drug

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. Known liver transplant or plan to transplant
3. GI hemorrhage with 6 months
4. History or current brain metastases
5. Active known, or suspected autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Haerbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - 81 Hospital Nanjing, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Zhangshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai

REFERENCES:
- [Derived] Zhou X, Cao J, Topatana W, Xie T, Chen T, Hu J, Li S, Juengpanic S, Lu Z, Zhang B, Wang K, Feng X, Shen J, Chen M. Evaluation of PD-L1 as a biomarker for immunotherapy for hepatocellular carcinoma: systematic review and meta-analysis. Immunotherapy. 2023 Apr;15(5):353-365. doi: 10.2217/imt-2022-0168. Epub 2023 Feb 27. PMID 36852452
- [Derived] Shi J, Liu J, Tu X, Li B, Tong Z, Wang T, Zheng Y, Shi H, Zeng X, Chen W, Yin W, Fang W. Single-cell immune signature for detecting early-stage HCC and early assessing anti-PD-1 immunotherapy efficacy. J Immunother Cancer. 2022 Jan;10(1):e003133. doi: 10.1136/jitc-2021-003133. PMID 35101942
- [Derived] Qin S, Ren Z, Meng Z, Chen Z, Chai X, Xiong J, Bai Y, Yang L, Zhu H, Fang W, Lin X, Chen X, Li E, Wang L, Chen C, Zou J. Camrelizumab in patients with previously treated advanced hepatocellular carcinoma: a multicentre, open-label, parallel-group, randomised, phase 2 trial. Lancet Oncol. 2020 Apr;21(4):571-580. doi: 10.1016/S1470-2045(20)30011-5. Epub 2020 Feb 26. PMID 32112738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
Started | 111 | 109
Treated | 109 | 108
Completed | 72 | 81
Not Completed | 39 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W | Total
Number analyzed (Participants) | 109 | 108 | 217
Age, Continuous [Median (Full Range); unit: years] | 48.0 [25 to 80] | 49.5 [23 to 76] | 49.0 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 98 | 98 | 196
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 109 | 108 | 217

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Tumour responses were evaluated by the independent review committee (IRC) according to RECIST 1.1.The primary endpoints were the proportion of patients with a IRC-assessed objective response (defined as the percentage of patients whose best overall response was confirmed complete or partial response).
Time Frame: approximate 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
Number analyzed (Participants) | 109 | 108
percentage of participants | 11.9 [6.5 to 19.5] | 16.7 [10.2 to 25.1]

2. Primary Outcome: 6-month Overall Survival Rate
Description: 6-month overall survival rate (defined as cumulative overall survival rate from the date of the first dose to 6 months)
Time Frame: from the date of the first dose to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
Number analyzed (Participants) | 109 | 108
percentage of participants | 75.9 [66.6 to 82.9] | 73.0 [63.6 to 80.4]

3. Secondary Outcome: Duration of Response
Description: time from first response to progression or death base on the IRC assessment
Time Frame: approximate 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
Number analyzed (Participants) | 109 | 108
months | 30.4 [2.8 to NA] — not reached (due to insufficient number of subjects with events). | 30.5 [5.4 to NA] — not reached (due to insufficient number of subjects with events).

4. Secondary Outcome: Adverse Events
Description: Number of Subjects with one or more adverse events as assessed by CTCAE 4.03
Time Frame: approximate 3 years
Measure: Number; unit: participants
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
Number analyzed (Participants) | 109 | 108
participants | 109 | 108

5. Secondary Outcome: Overall Survival
Description: Time from first dose to death from any cause
Time Frame: approximate 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
Number analyzed (Participants) | 109 | 108
months | 14.3 [11.5 to 19.5] | 13.2 [9.4 to 16.3]

ADVERSE EVENTS:
Time Frame: approximate 3 years
Description: Adverse events were monitored and recorded from the time of informed consent until 90 days after last administration and were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.
Arm/Group | SHR-1210 Q2W | SHR-1210 Q3W
All-Cause Mortality (participants affected / at risk) | 27/109 | 29/108
Serious Adverse Events (participants affected / at risk) | 50/109 | 46/108
Other Adverse Events (participants affected / at risk) | 108/109 | 107/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SHR-1210 Q2W (N=109) | SHR-1210 Q3W (N=108)
Disease progression (General disorders) | 13 | 9
Multiple organ dysfunction syndrome (General disorders) | 3 | 3
Death (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 6
Hepatic failure (Hepatobiliary disorders) | 4 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4
Ascites (Gastrointestinal disorders) | 1 | 1
Oral reactive capillary endothelial proliferation (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Splenic abscess (Infections and infestations) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Reactive cutaneous capillary endothelial proliferation (Skin and subcutaneous tissue disorders) | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0
Nasal mucosal reactive capillary endothelial proliferation (Vascular disorders) | 0 | 1
Vascular rupture (Vascular disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SHR-1210 Q2W (N=109) | SHR-1210 Q3W (N=108)
Anaemia (Blood and lymphatic system disorders) | 27 | 28
Hypothyroidism (Endocrine disorders) | 14 | 13
Hyperthyroidism (Endocrine disorders) | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 17 | 20
Abdominal distension (Gastrointestinal disorders) | 11 | 15
Ascites (Gastrointestinal disorders) | 12 | 13
Abdominal pain (Gastrointestinal disorders) | 11 | 10
Abdominal pain upper (Gastrointestinal disorders) | 7 | 13
Nausea (Gastrointestinal disorders) | 10 | 8
Constipation (Gastrointestinal disorders) | 5 | 6
Pyrexia (General disorders) | 26 | 23
Asthenia (General disorders) | 23 | 23
Oedema peripheral (General disorders) | 7 | 6
Chest pain (General disorders) | 7 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 10 | 15
Jaundice (Hepatobiliary disorders) | 3 | 9
Upper respiratory tract infection (Infections and infestations) | 17 | 12
Urinary tract infection (Infections and infestations) | 3 | 8
Aspartate aminotransferase increased (Investigations) | 52 | 48
Alanine aminotransferase increased (Investigations) | 47 | 46
Blood bilirubin increased (Investigations) | 40 | 38
Platelet count decreased (Investigations) | 35 | 39
White blood cell count decreased (Investigations) | 24 | 31
Neutrophil count decreased (Investigations) | 23 | 26
Weight increased (Investigations) | 27 | 21
Bilirubin conjugated increased (Investigations) | 25 | 20
Gamma-glutamyltransferase increased (Investigations) | 17 | 28
Blood alkaline phosphatase increased (Investigations) | 18 | 21
Weight decreased (Investigations) | 14 | 17
Blood albumin decreased (Investigations) | 13 | 11
Blood lactate dehydrogenase increased (Investigations) | 9 | 15
Lymphocyte count decreased (Investigations) | 10 | 13
Blood thyroid stimulating hormone increased (Investigations) | 11 | 10
Lipase increased (Investigations) | 7 | 12
Blood bilirubin unconjugated increased (Investigations) | 8 | 10
Hepatitis B DNA increased (Investigations) | 7 | 11
Protein urine present (Investigations) | 5 | 8
Neutrophil count increased (Investigations) | 2 | 8
White blood cell count increased (Investigations) | 1 | 9
Blood glucose increased (Investigations) | 6 | 3
Decreased appetite (Metabolism and nutrition disorders) | 22 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 18
Hypoproteinaemia (Metabolism and nutrition disorders) | 14 | 16
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 69 | 76
Headache (Nervous system disorders) | 9 | 4
Insomnia (Psychiatric disorders) | 3 | 6
Proteinuria (Renal and urinary disorders) | 36 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 13 | 12
Hypertension (Vascular disorders) | 18 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT02989922/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02989922/SAP_001.pdf